CLINICAL TRIAL: NCT01956617
Title: The Mininimum Effective Anaesthetic Volume of Local Anaesthetic in Ultrasound-guided "Shamrock" Lumbar Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Axel Rudolf Sauter, MD. PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: 2013/1328-3
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Mininimum Effective Anaesthetic Volume of Local Anaesthetic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- injection volume (Other): block success or failure determines a 5 ml decrease or increase for the subsequent patient, respectively
  Interventions: Other: lumbar plexus block

INTERVENTIONS:
Other: lumbar plexus block

SUMMARY:
The "Shamrock method" is a new ultrasound-guided lumbar plexus block. The aim of the study is to determine the minimum effective volume of ropivacaine 0.5% required to produce an effective lumbar plexus block with this method. Using the Dixon and Massey up-and-down method study design, 30 patients scheduled for elective total hip and knee arthroplasty will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* orthopaedic patients scheduled for elective hip and knee arthoroplasty
* ASA 1 - 2 or stable ASA 3
* age between 18 and 70 years
* good ability to communicate and to cooperate

Exclusion Criteria:

* ASA > 3 or unstable ASA 3
* BMI > 32
* chronicle pain
* nephrological diseases or nephropathy
* known contraindications against the use of local anaesthetics
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
minimum effective volume | from day 1 up to 20 weeks
  The primary outcome measure (MEV) is based on 30 measurements in 30 patients (secondary outcome measure: block success). MEV is determined by Dixon and Massey up-and-down method when all patients have been tested in the study

SECONDARY OUTCOMES:
block success | Day 1
  45 minutes after lumbar plexus blockade was performed

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Department of Anaesthesia and Intensive Care Medicine, Oslo University Hospital, Oslo, Oslo County
  - Oslo University Hospital, Oslo, Oslo County

REFERENCES:
- [Derived] Sauter AR, Ullensvang K, Niemi G, Lorentzen HT, Bendtsen TF, Borglum J, Pripp AH, Romundstad L. The Shamrock lumbar plexus block: A dose-finding study. Eur J Anaesthesiol. 2015 Nov;32(11):764-70. doi: 10.1097/EJA.0000000000000265. PMID 26426575